CLINICAL TRIAL: NCT05347082
Title: Resolution of Hyperparathyroidism With High-dose Vitamin D Improves Osteoporosis in Multi-treated Postmenopausal Women
Brief Title: Frequency of Hyperparathyroidism in Postmenopausal Osteoporosis and Its Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional 1o de Octubre (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120.2021
Record Dates: First submitted 2022-04-17; First posted 2022-04-26 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Postmenopausal Osteoporosis; Postmenopause; Hyperparathyroidism, Secondary; Hypovitaminosis D; Hyperparathyroidism, Primary
Keywords: Vitamin D; Postmenopause; Osteopenia; Osteoporosis; Bone Mineral Density; Hyperparathyroidism
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Hyperparathyroidism, Secondary; Vitamin D Deficiency; Hyperparathyroidism, Primary; Bone Diseases, Metabolic; Osteoporosis; Hyperparathyroidism | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: 47 participants who met the inclusion criteria were included and all received 8000 IU of vitamin D orally for four weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Experimental): 8000 IU of vitamin D orally, once a day, for four weeks.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Tablets of 4000 IU
  Other Names: Histofil®

SUMMARY:
Recently, an increase in the prevalence of hyperparathyroidism and hypovitaminosis D in postmenopause women has been occurring in Mexico and the world. Chronic exposure to the parathyroid hormone (PTH) is catabolic for the bone, worsening the state of osteoporosis. However, it is unclear whether these conditions could significantly improve bone mineral density (BMD). In the present work, it was shown that the resolution of hyperparathyroidism in postmenopausal women improves osteoporosis.

DETAILED DESCRIPTION:
This study was an open clinical trial conducted in Mexican women diagnosed with postmenopausal osteoporosis and hyperparathyroidism associated or not with hypovitaminosis D from the climacteric clinic of the regional hospital "1o de Octubre" of the Institute of Security and Social Services for State Workers (ISSSTE).

An integral clinical evaluation with PTH and vitamin D measurement was first done to determine the frequency of primary hyperparathyroidism and hypovitaminosis D. Likewise, a thyroid ultrasound was done. Then, 8000 IU of vitamin D were orally administrated for four weeks. Statical analysis was performed using PAST 3.0 and GraphPad Prism 8.4.3. software. The arithmetic median (µ) and standard deviation (S.D.) were calculated using Excel-Word. Graphics were constructed with GraphPad Prism 8.4.3 and tables with Excel-Word. Categorical variables were analysed with chi-squared or Fisher exact test depending on the number of participants in each cell. Normality was determined using the Shapiro-Wilk test. To compare two paired samples, the Wilcoxon signed-rank test was utilized. To perform correlations, the Spearman correlation coefficient was used. The assigned α value for this study was <0.05. In all cases, if a Montecarlo permutation was available, the exact p-value was taken instead of the raw p-value.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance to participate in the study with informed consent.
* Postmenopausal osteoporosis or osteopenia.
* Primary or secondary hyperparathyroidism.
* Insufficiency or deficiency of vitamin D.
* Multi-treated postmenopausal osteoporosis.
* Postmenopausal osteoporosis without treatment.

Exclusion Criteria:

* Different osteoporosis aetiology not related to oestrogenic deficiency.
* Thyroid pathology.
* Previous treatment with vitamin D, thiazide diuretics, lithium, Teriparatide or glucocorticoids.
* Known allergies to vitamin D.
* Addison's disease, pheochromocytoma, and depressive disorders.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Remission of Hyperparathyroidism | 4 weeks
  Clinical remission of hyperparathyroidism was evaluated after treatment.
Number of Participants with Remission of Hypovitaminosis D | 4 weeks.
  Clinical remission of vitamin D deficiency or insufficiency were evaluated after treatment.
Change from baseline hip T score at 4 weeks | 4 weeks
  Osteoporosis in the hip was determined by a T score greater than -2.5 and osteopenia was determined by a T score between -1 to -2.4.
Change from baseline lumbar spine T score at 4 weeks | 4 weeks
  Osteoporosis in the lumbar spine was determined by a T-score greater than -2.5 and osteopenia was determined by a T-score between -1 and -2.4.

SECONDARY OUTCOMES:
Change from baseline general T score at 4 weeks | 4 weeks
  Osteoporosis was determined by a T-score greater than -2.5 either in the hip or in the lumbar spine and osteopenia was determined by a T-score between -1 and -2.4 either in the hip or in the lumbar spine.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Ocampo Godínez, M.D., Ph.D., Study Director — Tissue Bioengineering Laboratory, National Autonomous University of Mexico [UNAM]; Patricia Loranca-Moreno, M.D., M.Sc., Study Director — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE.; Paula M Sánchez-Tinoco, M.D., Principal Investigator — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE.
Locations (1):
- Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosman F, de Beur SJ, LeBoff MS, Lewiecki EM, Tanner B, Randall S, Lindsay R; National Osteoporosis Foundation. Clinician's Guide to Prevention and Treatment of Osteoporosis. Osteoporos Int. 2014 Oct;25(10):2359-81. doi: 10.1007/s00198-014-2794-2. Epub 2014 Aug 15. PMID 25182228
- [Background] Lundgren E, Hagstrom EG, Lundin J, Winnerback K, Roos J, Ljunghall S, Rastad J. Primary hyperparathyroidism revisited in menopausal women with serum calcium in the upper normal range at population-based screening 8 years ago. World J Surg. 2002 Aug;26(8):931-6. doi: 10.1007/s00268-002-6621-0. Epub 2002 Jun 6. PMID 12045863
- [Background] Grey A, Lucas J, Horne A, Gamble G, Davidson JS, Reid IR. Vitamin D repletion in patients with primary hyperparathyroidism and coexistent vitamin D insufficiency. J Clin Endocrinol Metab. 2005 Apr;90(4):2122-6. doi: 10.1210/jc.2004-1772. Epub 2005 Jan 11. PMID 15644400
- [Background] Tucci JR. Vitamin D therapy in patients with primary hyperparathyroidism and hypovitaminosis D. Eur J Endocrinol. 2009 Jul;161(1):189-93. doi: 10.1530/EJE-08-0901. Epub 2009 Apr 21. PMID 19383807
- [Background] Contreras-Manzano A, Villalpando S, Robledo-Perez R. Vitamin D status by sociodemographic factors and body mass index in Mexican women at reproductive age. Salud Publica Mex. 2017 Sep-Oct;59(5):518-525. doi: 10.21149/8080. PMID 29267648
- [Background] Goltzman D. Functions of vitamin D in bone. Histochem Cell Biol. 2018 Apr;149(4):305-312. doi: 10.1007/s00418-018-1648-y. Epub 2018 Feb 12. PMID 29435763
- [Background] Lips P, van Schoor NM. The effect of vitamin D on bone and osteoporosis. Best Pract Res Clin Endocrinol Metab. 2011 Aug;25(4):585-91. doi: 10.1016/j.beem.2011.05.002. PMID 21872800
- [Background] Lips P. Vitamin D deficiency and secondary hyperparathyroidism in the elderly: consequences for bone loss and fractures and therapeutic implications. Endocr Rev. 2001 Aug;22(4):477-501. doi: 10.1210/edrv.22.4.0437. PMID 11493580
- [Background] Recker RR, Kendler D, Recknor CP, Rooney TW, Lewiecki EM, Utian WH, Cauley JA, Lorraine J, Qu Y, Kulkarni PM, Gaich CL, Wong M, Plouffe L Jr, Stock JL. Comparative effects of raloxifene and alendronate on fracture outcomes in postmenopausal women with low bone mass. Bone. 2007 Apr;40(4):843-51. doi: 10.1016/j.bone.2006.11.001. Epub 2006 Dec 19. PMID 17182297
- [Background] Manson JE, Hsia J, Johnson KC, Rossouw JE, Assaf AR, Lasser NL, Trevisan M, Black HR, Heckbert SR, Detrano R, Strickland OL, Wong ND, Crouse JR, Stein E, Cushman M; Women's Health Initiative Investigators. Estrogen plus progestin and the risk of coronary heart disease. N Engl J Med. 2003 Aug 7;349(6):523-34. doi: 10.1056/NEJMoa030808. PMID 12904517
- [Background] Watson J, Wise L, Green J. Prescribing of hormone therapy for menopause, tibolone, and bisphosphonates in women in the UK between 1991 and 2005. Eur J Clin Pharmacol. 2007 Sep;63(9):843-9. doi: 10.1007/s00228-007-0320-6. Epub 2007 Jun 28. PMID 17598097
- [Background] Davis S, Martyn-St James M, Sanderson J, Stevens J, Goka E, Rawdin A, Sadler S, Wong R, Campbell F, Stevenson M, Strong M, Selby P, Gittoes N. A systematic review and economic evaluation of bisphosphonates for the prevention of fragility fractures. Health Technol Assess. 2016 Oct;20(78):1-406. doi: 10.3310/hta20780. PMID 27801641
- [Background] Paggiosi MA, Peel N, McCloskey E, Walsh JS, Eastell R. Comparison of the effects of three oral bisphosphonate therapies on the peripheral skeleton in postmenopausal osteoporosis: the TRIO study. Osteoporos Int. 2014 Dec;25(12):2729-41. doi: 10.1007/s00198-014-2817-z. Epub 2014 Jul 30. PMID 25074351
- [Background] Chen LX, Zhou ZR, Li YL, Ning GZ, Zhang TS, Zhang D, Feng SQ. Comparison of Bone Mineral Density in Lumbar Spine and Fracture Rate among Eight Drugs in Treatments of Osteoporosis in Men: A Network Meta-Analysis. PLoS One. 2015 May 26;10(5):e0128032. doi: 10.1371/journal.pone.0128032. eCollection 2015. PMID 26010450
- [Background] Yuan F, Peng W, Yang C, Zheng J. Teriparatide versus bisphosphonates for treatment of postmenopausal osteoporosis: A meta-analysis. Int J Surg. 2019 Jun;66:1-11. doi: 10.1016/j.ijsu.2019.03.004. Epub 2019 Mar 16. PMID 30890377
- [Background] Chang B, Quan Q, Li Y, Qiu H, Peng J, Gu Y. Treatment of Osteoporosis, with a Focus on 2 Monoclonal Antibodies. Med Sci Monit. 2018 Dec 3;24:8758-8766. doi: 10.12659/MSM.912309. PMID 30508820
- [Background] Leder BZ, Tsai JN, Uihlein AV, Wallace PM, Lee H, Neer RM, Burnett-Bowie SA. Denosumab and teriparatide transitions in postmenopausal osteoporosis (the DATA-Switch study): extension of a randomised controlled trial. Lancet. 2015 Sep 19;386(9999):1147-55. doi: 10.1016/S0140-6736(15)61120-5. Epub 2015 Jul 2. PMID 26144908
- [Background] Lundgren E, Rastad J, Thrufjell E, Akerstrom G, Ljunghall S. Population-based screening for primary hyperparathyroidism with serum calcium and parathyroid hormone values in menopausal women. Surgery. 1997 Mar;121(3):287-94. doi: 10.1016/s0039-6060(97)90357-3. PMID 9092129
- [Background] Wihlborg A, Bergstrom K, Gerdhem P, Bergstrom I. Parathyroid Hormone Disturbances in Postmenopausal Women with Distal Forearm Fracture. World J Surg. 2022 Jan;46(1):128-135. doi: 10.1007/s00268-021-06331-w. Epub 2021 Oct 13. PMID 34647149
- [Background] Souberbielle JC, Bienaime F, Cavalier E, Cormier C. Vitamin D and primary hyperparathyroidism (PHPT). Ann Endocrinol (Paris). 2012 Jun;73(3):165-9. doi: 10.1016/j.ando.2012.04.008. Epub 2012 Jun 5. PMID 22677209
- [Background] Rolighed L, Rejnmark L, Sikjaer T, Heickendorff L, Vestergaard P, Mosekilde L, Christiansen P. Vitamin D treatment in primary hyperparathyroidism: a randomized placebo controlled trial. J Clin Endocrinol Metab. 2014 Mar;99(3):1072-80. doi: 10.1210/jc.2013-3978. Epub 2014 Jan 13. PMID 24423366
- [Background] Holick MF, Siris ES, Binkley N, Beard MK, Khan A, Katzer JT, Petruschke RA, Chen E, de Papp AE. Prevalence of Vitamin D inadequacy among postmenopausal North American women receiving osteoporosis therapy. J Clin Endocrinol Metab. 2005 Jun;90(6):3215-24. doi: 10.1210/jc.2004-2364. Epub 2005 Mar 29. PMID 15797954
- [Background] Neuprez A, Bruyere O, Collette J, Reginster JY. Vitamin D inadequacy in Belgian postmenopausal osteoporotic women. BMC Public Health. 2007 Apr 26;7:64. doi: 10.1186/1471-2458-7-64. PMID 17462085